CLINICAL TRIAL: NCT05907850
Title: A Randomized Placebo-controlled Trial Investigating the Effects of Riboflavin in Mitigating Muscle Soreness in Ultra-marathon Athletes
Brief Title: Effects of Riboflavin in Mitigating Muscle Soreness in Ultra-marathon Athletes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Steven Moore (Other)
Collaborators: Racing the Planet (Unknown)
Responsible Party: Sponsor-Investigator, Steven Moore, Associate Professor, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20230413H
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Muscle Soreness
Keywords: Delayed onset muscle soreness; Ultramarathon
MeSH Terms: conditions — Myalgia | interventions — Riboflavin

STUDY DESIGN:
Intervention Model Description: A phase I randomized, 2 arm single blinded feasibility study
Who Masked: Participant
Masking Description: Subjects will be masked to which intervention they receive, active study drug or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riboflavin Group (Active Comparator): Riboflavin 100mg will be self administered by participants, one capsules prior to the long stage of the race followed by a second dose at the completion of the long stage.
  Interventions: Drug: Riboflavin
- Placebo/Control Group (Placebo Comparator): Placebo will be self administered by participants, one capsule prior to the long stage of the race followed by a second dose at the completion of the long stage.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riboflavin — Commercially available source of riboflavin capsules
  Other Names: Riboflavin 100mg capsules
  Arms: Riboflavin Group
Drug: Placebo — Placebo capsule compounded to be similar in appearance to the active intervention
  Other Names: Placebo capsule
  Arms: Placebo/Control Group

SUMMARY:
The aim of this project is to investigate the effects of riboflavin, also known as vitamin B2, on preventing delayed onset muscle soreness (DOMS) in ultramarathon athletes through a randomized placebo-controlled study.

DETAILED DESCRIPTION:
The riboflavin 100 mg capsules will be self-dosed by the participant, one capsule prior to the long stage of the race followed by a second dose at the end of the long stage. Historically, long-stage finish times have ranged between 8 and 24 hours. The placebo will also be dosed as one capsule on the morning of the long stage, prior to the race start, and one capsule at the end of the long stage.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or over
4. In good general health as evidenced by readiness to participate in an ultramarathon
5. Ability to take oral medication and be willing to adhere to the study regimen
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening.

Exclusion Criteria:

1. Unable to read or understand English
2. Under 18 years of age
3. Pregnancy or lactation
4. Known allergic reactions to components of the investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Muscle soreness measure for long stage of the ultramarathon | Baseline to 6 days
  Change in muscle soreness at completion of the long stage (80+ kilometers) of the ultramarathon. Muscle soreness the day following long stage completion. Muscle soreness will be measured using a Likert scale rated from 0 to 10 where 0 indicates no soreness and 10 indicates unbearable pain.

SECONDARY OUTCOMES:
Muscle soreness measure post-race | Day 7
  Muscle soreness the day following long stage completion. Muscle soreness the day following long stage completion. Muscle soreness will be measured using a Likert scale rated from 0 to 10 where 0 indicates no soreness and 10 indicates unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Moore, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States